CLINICAL TRIAL: NCT07142122
Title: Safety Comparison of Total Laparoscopic Proximal Gastrectomy With or Without Preservation of the Celiac Branch of the Vagus Nerve for Early Upper Gastric Cancer: A Randomized Controlled Clinical Trial
Acronym: TLPG-CBVP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLPG-CBVP; 2023-2839 (Other Grant/Funding Number: Fujian Provincial Young and Middle-aged Health Leading Talent Training Program)
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Gastric Cancer
Keywords: Esophagogastric Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Group A) (Experimental): Total laparoscopic proximal gastrectomy with preservation of hepatic and celiac branches of the vagus nerve. Reconstruction by double-tract anastomosis.
  Interventions: Procedure: Total laparoscopic proximal gastrectomy with preservation of both the hepatic and celiac branches of the vagus nerve, followed by double-tract reconstruction.
- Active Comparator Arm (Group B) (Active Comparator): Procedure: Total laparoscopic proximal gastrectomy with preservation of hepatic branch but without preservation of the celiac branch of the vagus nerve. Reconstruction by double-tract anastomosis.
  Interventions: Procedure: Total laparoscopic proximal gastrectomy with preservation of the hepatic branch of the vagus nerve but deliberate resection of the celiac branch, followed by double-tract reconstruction.

INTERVENTIONS:
Procedure: Total laparoscopic proximal gastrectomy with preservation of both the hepatic and celiac branches of the vagus nerve, followed by double-tract reconstruction. — Total laparoscopic proximal gastrectomy with meticulous preservation of the hepatic branch of the vagus nerve (via fenestration of the lesser omentum) and the celiac branch (via skeletonization of the left gastric artery). The esophagus was transected ≥3 cm proximal to the tumor, preserving >50% of the residual stomach. Double-tract reconstruction was then performed: an end-to-side esophagojejunostomy was created first, followed by a side-to-side gastrojejunostomy between the residual stomach and jejunum, and finally a side-to-side jejunojejunostomy approximately 40 cm distal to the gastrojejunal anastomosis. This approach achieves oncological resection while maximizing preservation of digestive physiology (gallbladder contraction, reduced dumping syndrome, and partial gastric reservoir function).
  Arms: Experimental Arm (Group A)
Procedure: Total laparoscopic proximal gastrectomy with preservation of the hepatic branch of the vagus nerve but deliberate resection of the celiac branch, followed by double-tract reconstruction. — Total laparoscopic proximal gastrectomy with meticulous preservation of the hepatic branch of the vagus nerve (via lesser omentum fenestration adjacent to the liver edge), while deliberately not preserving the celiac branch (by direct transection at the root of the left gastric artery). The esophagus was transected ≥3 cm proximal to the tumor with preservation of >50% gastric remnant. Double-tract reconstruction was then executed: end-to-side esophagojejunostomy (circular stapler) → side-to-side gastrojejunostomy (linear cutter) → side-to-side jejunojejunostomy approximately 40 cm distal to the gastrojejunal anastomosis. This technique achieves oncological resection while utilizing the residual stomach and dual-pathway design to minimize postoperative dumping syndrome and preserve partial gastric function.
  Arms: Active Comparator Arm (Group B)

SUMMARY:
This prospective, single-center, randomized, controlled, non-inferiority clinical trial aims to compare the safety and postoperative quality of life of early upper gastric cancer patients undergoing total laparoscopic proximal gastrectomy (TLPG) with preservation of both the hepatic and celiac branches of the vagus nerve versus preservation of the hepatic branch only. The primary endpoint is gastric emptying half-time of solid food at 6 months after surgery. Secondary outcomes include incidence of reflux esophagitis, quality of life scores (EORTC QLQ-C30/STO22), number and positivity rate of lymph nodes retrieved, and 3-year disease-free survival. The study will provide evidence for optimizing minimally invasive surgical strategies for early upper gastric cancer.

DETAILED DESCRIPTION:
Early gastric cancer involving the upper third of the stomach or esophagogastric junction is increasingly managed with minimally invasive surgery. The vagus nerve plays an essential role in regulating gastric motility and postoperative physiological recovery. Preservation of the hepatic branch is widely accepted, while the role of preserving the celiac branch remains controversial. This trial is designed to evaluate whether preservation of the celiac branch during TLPG improves gastric emptying and postoperative quality of life without compromising oncological safety. Eligible patients (cT1bN0M0, tumor size ≤4 cm, no prior chemotherapy/radiotherapy) will be randomized into two groups: Group A (hepatic and celiac branches preserved) and Group B (hepatic branch preserved only). Both groups undergo double-tract reconstruction. The study will enroll 76 patients (38 per group) with sufficient statistical power. Outcomes will be analyzed using standard statistical methods, and the findings are expected to provide evidence for refined vagus-nerve-preserving surgery in early gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Histologically confirmed gastric adenocarcinoma or esophagogastric junction adenocarcinoma (papillary, tubular, mucinous, poorly cohesive including signet-ring cell carcinoma, or mixed type).
3. Primary tumor located in the upper third of the stomach, or esophagogastric junction cancer with tumor size ≤4 cm.
4. Clinical stage cT1bN0M0 without lymph node metastasis.
5. BMI <30 kg/m².
6. No history of upper abdominal surgery (except laparoscopic cholecystectomy).
7. No prior chemotherapy, radiotherapy, targeted therapy, or immunotherapy.
8. ECOG performance status 0-1.
9. ASA class I-III.
10. Adequate organ function.
11. Signed informed consent.

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Other malignancies within 5 years.
3. Active infection requiring systemic therapy or fever ≥38°C preoperatively.
4. Severe psychiatric illness.
5. Severe respiratory disease.
6. Severe hepatic or renal dysfunction.
7. Unstable angina or myocardial infarction within 6 months.
8. Stroke or intracranial hemorrhage within 6 months.
9. Long-term systemic glucocorticoid therapy within 1 month (local use excluded).
10. Complications of gastric cancer (bleeding, perforation, obstruction).
11. Participation in another clinical study within 6 months.

Exclusion During Study (Removal Criteria):

R0 resection not achieved, change of procedure to total gastrectomy or PPG, combined surgery for other diseases, severe perioperative complications, emergency surgery required, patient withdrawal of consent, or protocol violation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Gastric half-emptying time of solid food at 6 months postoperatively (minutes, measured by gastric emptying test) | 6 months post-operation

SECONDARY OUTCOMES:
Reflux Esophagitis (LA Classification) | 1,3,6,12,24 months
EORTC QLQ-C30/STO22 Scores | 1,3,6,12,24 months
Lymph Node Yield/Positivity Rate | Intraoperative
3-Year Disease-Free Survival | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- 420 Fuma Road, Jin'an District, Fuzhou City, Fujian Province, Fuzhou, Fujian, China